CLINICAL TRIAL: NCT03831854
Title: The Role of Lamotrigine in Reducing Psychologic Side-Effect of Perioperative Ketamine Use
Brief Title: Lamotrigine in Reducing Psychologic Side-Effect of Perioperative Ketamine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 18-952
Record Dates: First submitted 2018-12-03; First posted 2019-02-06 (Actual); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Reducing Psychological Side Effects of Ketamine
MeSH Terms: interventions — Lamotrigine; Ketamine

STUDY DESIGN:
Intervention Model Description: randomization without stratification
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Pharmacy will know the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- lamotrigine (Active Comparator): Patient will receive 300 mg of oral lamotrigine with small sips of water to reduce the psychologic side effects (measured by four key items of Brief Psychiatric Rating Scale: conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content) of intraoperative ketamine use.
  Interventions: Drug: Lamotrigine 300 MG; Drug: Ketamine
- Placebo (Placebo Comparator): Patient will receive oral Placebo with small sips of water, to reduce the psychologic side effects (measured by four key items of Brief Psychiatric Rating Scale: conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content) of intraoperative ketamine use.
  Interventions: Drug: Placebo; Drug: Ketamine

INTERVENTIONS:
Drug: Lamotrigine 300 MG — 300 mg of oral Lamotrigine. One of the key studies in this area was reported at the Society of Neuroscience meeting in 1997 and later published in the Archives of General Psychiatry. This study reported that, in healthy subjects 300 mg oral lamotrigine significantly decreased ketamine-induced perceptual abnormalities as assessed by the Clinician-Administered Dissociative States Scale (P<.001).31 Furthermore lamotrigine increased the immediate mood-elevating effects of ketamine (P<.05).
  Other Names: Lamictal 300 mg
  Arms: lamotrigine
Drug: Placebo — 300 mg of oral Placebo
  Arms: Placebo
Drug: Ketamine — 1mg/kg bolus at induction followed by 5 microgram/kg/min infusion till the end of the surgery

SUMMARY:
Patient will receive lamotrigine vs. placebo with small sips of water. Lamotrigine reaches peak level 1-4 hours after oral administration.

DETAILED DESCRIPTION:
1:1 randomization without stratification use web-based software (Redcap) before surgery. Allocation will be concealed from the patient, the nurse, the operating room team. Both patient and the operating room team will be blinded to the treatment allocation (double blind).

Standard preoperative care as per anesthesia care team. Patient will receive lamotrigine vs. placebo with small sips of water. Lamotrigine reaches peak level 1-4 hours after oral administration. Single dose lamotrigine is safe and is not associated with rash.

Standard intraoperative care as per the anesthesia care team. All patients will receive Ketamine 1 mg/kg at induction. Ketamine 5mcg/kg/min will be started at induction and stopped at the end of surgery.

Standard postoperative care as per PACU team. The psychologic side-effects will be measured using Brief Psychiatric Rating Scale (BPRS) using an online tool.

Research fellow will receive standardized training in administering BPRS from Dr. Amit Anand using structured material. Dr. Anand has used this training for other current research projects.

ELIGIBILITY:
Inclusion Criteria:

* 18 -65 Years of age
* Planned overnight hospital stay

Exclusion Criteria:

* Pregnant and planning to become pregnant
* No known History of seizure
* No known History of Schizophrenia
* No known History of unstable angina
* Patients taking Antiepileptic medications
* Known history of Lamotrigine intake in past.
* Any history of allergic reaction to lamotrigine in the past.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make subjects data available to outside researchers

RESULTS

PARTICIPANT FLOW:
Groups:
- Lamotrigine: Preoperatively, the patient will receive 300 mg of oral lamotrigine pill with small sips of water once.
- Placebo: Preoperatively, the patient will receive a 300 mg oral placebo pill with small sips of water once.
Period: Overall Study
Arm/Group | Lamotrigine | Placebo
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamotrigine | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (13) | 42 (12) | 43 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 12 | 9 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 19 | 39
  Other | 3 | 4 | 7
ASA status, No (%) [Count of Participants; unit: Participants] — The ASA Physical Status Classification System is to assess and communicate a patient's pre-anesthesia medical co-morbidities. ASA scores included I, II, III, IV, V, and VI where I means normal status (best) and VI means a declared brain-dead patient whose organs are being removed for donor purposes (worst).
  Participants
    I | 1 | 0 | 1
    II | 9 | 12 | 21
    III | 13 | 11 | 24
History of alcoholism [Count of Participants; unit: Participants] | 3 | 2 | 5
Surgery duration (hours) [Median (Inter-Quartile Range); unit: hours] | 4 [3 to 5] | 3 [2 to 5] | 3.5 [3 to 5]
Surgery type [Count of Participants; unit: Participants]
  Orthopedic | 2 | 2 | 4
  Abdominal | 20 | 17 | 37
  General | 1 | 4 | 5
Hypertension [Count of Participants; unit: Participants] | 4 | 5 | 9
Chronic pulmonary disease [Count of Participants; unit: Participants] | 2 | 0 | 2
Diabetes [Count of Participants; unit: Participants] | 1 | 0 | 1
Renal failure [Count of Participants; unit: Participants] | 0 | 0 | 0
Psychoses [Count of Participants; unit: Participants] | 0 | 0 | 0
Depression [Count of Participants; unit: Participants] | 4 | 5 | 9
Other neurological disorders [Count of Participants; unit: Participants] | 1 | 0 | 1
BPRS(Brief Psychiatric Rating Scale) baseline score [Median (Inter-Quartile Range); unit: scores] — Brief Psychiatric Rating Scale (BPRS) corresponding to positive symptoms of schizophrenia: conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content. Each symptom is rated 1-7 ( 1 = not present, 2 = very mild, 3 = mild, 4 = moderate, 5 = moderately severe, 6 = severe, 7 = extremely severe ), and, therefore, the total score based on four key items of BPRS will be between 4 (best score) and 28 (worst score).
  scores | 25 [25 to 27] | 25 [24 to 27] | 25 [24 to 27]
Positive symptoms of schizophrenia based on four key items of BPRS (Brief Psychiatric Rati)-baseline [Count of Participants; unit: Participants] | 1 | 2 | 3
Total dose of Ketamine, mg [Mean (Standard Deviation); unit: mg] | 143 (48) | 142 (54) | 143 (51)

OUTCOME MEASURES:

1. Primary Outcome: Psychologic Side-effects
Description: The primary outcome of psychologic side-effects was measured in PACU (up to 90 minutes after ketamine infusion). This included four key items of the Brief Psychiatric Rating Scale (BPRS) corresponding to positive symptoms of schizophrenia: conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content. Each symptom is rated 1-7 ( 1 = not present, 2 = very mild, 3 = mild, 4 = moderate, 5 = moderately severe, 6 = severe, 7 = extremely severe ), and, therefore, the total score as the primary outcome based on four key items of BPRS will be between 4 (best score) and 28 (worst score).
Time Frame: in PACU (up to 90 minutes after ketamine infusion)
Population: 46 patients were analyzed but 3 people were missing on the primary outcome.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 22 | 21
score on a scale | 4 [4 to 4] | 4 [4 to 4]
Statistical Analysis 1: Comparison: Lamotrigine vs Placebo; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0]

2. Primary Outcome: Number of Patients With Psychologic Disturbances-
Description: The psychologic side-effects were measured in PACU (up to 90 minutes after ketamine infusion). This included four key items of the Brief Psychiatric Rating Scale (BPRS) corresponding to positive symptoms of schizophrenia: conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content. Each symptom is rated 1-7 ( 1 = not present, 2 = very mild, 3 = mild, 4 = moderate, 5 = moderately severe, 6 = severe, 7 = extremely severe ), and, therefore, the total score as the primary outcome based on four key items of BPRS will be between 4 (best score) and 28 (worst score). Patients who had a total score of 4 (all symptoms not present) were determined as not having psychologic disturbance and patients who had a total score of > 4 (having any symptoms present) were determined as having psychologic disturbance.
Time Frame: Up to 90 minutes of PACU arrival
Population: A total of 3 people were missing on this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 22 | 21
Participants | 0 | 3
Statistical Analysis 1: Comparison: Lamotrigine vs Placebo; Test type: Superiority; p = 0.11, Fisher Exact; The relative risk could not be assessed due to zero incidence in the treatment group

3. Secondary Outcome: Total Opioid Consumption in PACU (mg)
Description: Total cumulative opioid use (total IV morphine equivalents) in postoperative anesthesia care unit (PACU)
Time Frame: from entry to PACU to leaving PACU, up to 4 hours
Population: The final study population.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 23 | 23
mg | 5 [0 to 15] | 10 [0 to 15]
Statistical Analysis 1: Comparison: Lamotrigine vs Placebo; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -2.3, 98.5% CI 2-sided [-9.5 to 5.0]

4. Secondary Outcome: Pain Score in PACU
Description: Pain score was scaled from 0-10 where 0 means no pain and 10 means most pain. The time-weighted average of pain scores was used if the pain score was measured multiple times.
Time Frame: from entry to PACU to leaving PACU
Population: The final study population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 23 | 23
score on a scale | 4.9 (3.1) | 4.4 (2.8)
Statistical Analysis 1: Comparison: Lamotrigine vs Placebo; Test type: Superiority; p = 0.58, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 98.3% CI 2-sided [-1.7 to 2.6]

5. Secondary Outcome: Number of Patients Who Had PONV (Postoperative Nausea Vomiting)
Description: PONV was measured through Postoperative Nursing Progress Record, where nausea vomiting severity was recorded as 0 (none), 1 (mild), 2 (moderate), 3 (severe). Patients whose score was 0 were determined as not having PONV and patients whose score was positive were determined as having PONV.
Time Frame: after surgery up to discharge
Population: Two patients were missing on this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 22 | 22
Participants | 5 | 5
Statistical Analysis 1: Comparison: Lamotrigine vs Placebo; Test type: Superiority; p = 1.0, Chi-squared; Risk Ratio (RR) = 1.0, 98.3% CI 2-sided [0.3 to 3.8]

6. Other Pre Specified Outcome: Daily Average Opioid Use During Hospital Stay
Description: The average daily opioid use (mg) during the hospital stay.
Time Frame: from admission up to discharge
Population: The final study population.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 23 | 23
mg | 24 [15 to 69] | 24 [15 to 58]

7. Other Pre Specified Outcome: Opioid Related Side-effects (ORSDS)-POD1
Description: ORSDS is a 4 point-scale that evaluates 3 symptom distress dimensions (frequency, severity, bothersomeness for 12 opioid-related side effects, with a score of each item ranging from 0 to 4 where higher scores mean more side effects). The final ORSDS score is the average of all 12 scores from those 12 items, ranging from 0 to 4 where a higher score means worse outcome. This one measure ORSDS at postoperative day 1
Time Frame: postoperative day 1
Population: The final study population.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 23 | 23
score on a scale | 0.38 [0 to 0.58] | 0.57 [0 to 0.74]

8. Other Pre Specified Outcome: Opioid Related Side-effects (ORSDS)-POD2
Description: ORSDS is a 4 point-scale that evaluates 3 symptom distress dimensions (frequency, severity, bothersomeness for 12 opioid-related side effects, with a score of each item ranging from 0 to 4 where higher scores mean more side effects). The final ORSDS score is the average of all 12 scores from those 12 items, ranging from 0 to 4 where a higher score means a worse outcome. This one measure ORSDS at postoperative day 2.
Time Frame: postoperative day 2
Population: the final study population.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 23 | 23
score on a scale | 0.18 [0 to 3.5] | 0.26 [0.16 to 0.67]

9. Other Pre Specified Outcome: PACU Length of Stay, Hours
Description: Hours spent in PACU (Postanesthesia Care Unit).
Time Frame: in PACU
Population: the final study population
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 23 | 23
hours | 1 [1 to 1] | 2 [1 to 2]

ADVERSE EVENTS:
Time Frame: from the beginning of the study to discharge, up to 10 days.
Arm/Group | Lamotrigine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT03831854/Prot_SAP_000.pdf